CLINICAL TRIAL: NCT05149508
Title: Intraperitoneal Pressure Measurements in Children: a Retrospective Study
Brief Title: Intraperitoneal Pressure Measurements in Children
Acronym: IPM
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8412
Record Dates: First submitted 2021-11-24; First posted 2021-12-08 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2021-11

CONDITIONS: Peritoneal Dialysis
Keywords: Peritoneal Dialysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pediatric peritoneal dialysis is prescribed according to the type of dialysis, the volume infused and the dialysis time. The measurement of intraperitoneal pressure (IPP) is an important and easy indicator to perform. A IPP greater than 18 cmH20 has been correlated with pain and dyspnea, a IPP greater than 14 has been correlated with a higher risk of peritonitis and a IPP greater than 13 was correlated with higher mortality and a switch on hemodialysis. These data suggest the importance of routine IPP measurement. Few data are available in the pediatric population.

ELIGIBILITY:
Inclusion criteria:

* Minor subject (<18 years old)
* In stable peritoneal dialysis for more than 3 months
* Subject having had at least 3 IPP measurements
* At least 3 months after surgery to insert a peritoneal dialysis catheter
* Subject (and / or his parental authority) not having expressed, after being informed, his opposition to the reuse of his data for the purposes of this research.

Exclusion criteria:

- -Subject (or his parents) having expressed his (their) opposition to participating in the stud

Max Age: 17 Years | Sex: All
Age Groups: Child
Study Population: Minor subject (<18 years old) in stable peritoneal dialysis for more than 3 months and having had at least 3 IPP measurements
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2021-09-23 (Actual); Primary Completion 2022-03-23 (Actual); Study Completion 2022-03-23 (Actual)

PRIMARY OUTCOMES:
Study of good prescribing practices in children followed by peritoneal dialysis at Strasbourg University Hospital, by intraperitoneal pressure measurements | Files analysed retrospectively from January 01, 2001 to August 31, 2019 will be examined]

CONTACTS AND LOCATIONS:
Locations (1):
- Service : Pédiatrie 1 - Hôpitaux Universitaires de Strasbourg, Strasbourg, France